CLINICAL TRIAL: NCT06324409
Title: Increasing Access to Colorectal Cancer Screening Among Immigrants
Brief Title: ImmigrantScreen Telephone Reminder Trial in Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-350
Record Dates: First submitted 2024-03-05; First posted 2024-03-22 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Cancer Colorectal
Keywords: colorectal cancer screening; immigrant; participation; intervention; reminder; information
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: There is an intervention group and a comparison group in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reminder telephone call (Active Comparator): A reminder telephone call with information on colorectal cancer screening in the language of origin (Urdu or Somali) in addition to the reminder letter in Norwegian (usual care)
  Interventions: Behavioral: Reminder telephone call
- Comparison (No Intervention): The reminder letter in Norwegian (usual care) only

INTERVENTIONS:
Behavioral: Reminder telephone call — A reminder telephone call with information on colorectal cancer screening in the language of origin (Urdu or Somali) in addition to the reminder letter in Norwegian (usual care)
  Arms: Reminder telephone call

SUMMARY:
The goal of this randomized trial is to test the effect of a reminder telephone call in the official native language in the country where the invitee is born, in addition to the reminder letter in Norwegian on participation in the National Colorectal Cancer Screening Program in Pakistani and Somalian immigrants, compared to the reminder letter in Norwegian only.

The main question it aims to answer is:

•Does a reminder telephone call in the language of origin increase participation in colorectal cancer screening in Pakistani and Somalian immigrants in Norway?

Participants in this trial are individuals with Pakistan or Somalia as their country of birth invited to the National Colorectal Cancer Screening Program, who have not participated by mailing a faecal sample to the screening laboratory.

In the intervention group, the participants will be called in the official language in their country of origin, to inform about colorectal cancer screening, in addition to the reminder letter in Norwegian language sent to all non-participants.

Participants in the comparison group will only be sent the reminder letter in Norwegian language.

The researchers will compare differences in the participation rate in the National Colorectal Cancer Screening Program between the intervention and comparison groups.

DETAILED DESCRIPTION:
The aim of the project is to study the effect of reminding non-participant Somalian and Pakistani immigrant groups by a telephone call in the official native language in the country of birth, in addition to the reminder letter in Norwegian, by running a randomized trial. The outcome is participation in the National Colorectal Cancer Screening Program by taking a faecal sample with a mailed test kit.

The design of the trial is a parallel two-arm intervention study, with 1:1 randomization to intervention or control.

The intervention consists of a reminder both as telephone call in the native language of the non-participant's country of birth and the standard reminder letter (sent digitally or in mail) in Norwegian from the National Colorectal Cancer Screening Program. The timepoint of the telephone call will be during a week after the reminder letter has been mailed to the non-participant. The information to be given in the reminder call will include the same information as given in the reminder letter, but it will be asked additionally whether the invitee has understood the invitation and whether he/she has any questions. A new faecal sample kit will be sent on request.

The control arm will consist of screening practice as usual, which is the standard reminder letter in Norwegian from the National Colorectal Cancer Screening Program. A new faecal sample kit will be sent on request.

Masking: There is no masking in the trial. Allocation: This is a randomized trial. Participants are assigned to intervention groups by chance, using Random Integer Generator in random.org, when being assigned to the list of persons to whom a reminder is sent to.

Participation rate in the National Colorectal Cancer Screening Program will be compared between the intervention and control arms. That is, comparison of the proportion of individuals who send a faecal sample in mail to the screening laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Pakistan or Somalia registered as country of birth
* Invited to the first round of faecal screening test in the National Colorectal Cancer Screening Program in Norway
* Reminder letter sent after no received faecal sample in the screening laboratory within six weeks from mailing of the faecal screening sample kit from the screening organizers

Exclusion Criteria:

* Individuals whose mailed reminder letter is returned to sender
* Individuals whose faecal screening sample is registered in the screening laboratory 1) on the same day or the day after the reminder letter is sent out (applies to those who receive a digital reminder), or 2) on the same day or up to three days after the reminder letter is sent out (applies to those who receive a mailed reminder letter)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
First round screening participation | within 12 weeks (84 days) from mailing of the screening reminder letter
  Participation rate in the first colorectal cancer screening round. For each randomized individual, it is measured whether or not the faecal sample is sent to the screening laboratory by the participant in the first round of screening (yes/no).

SECONDARY OUTCOMES:
Overall screening participation | within six months from mailing of the last screening round invitation (of up to five rounds)
  Participation rate in all five rounds of colorectal cancer screening. For each randomized individual, it is measured to which degree faecal samples are sent to the screening laboratory by the participant (yes, in all five rounds of screening/yes, in 1-4 rounds of screening/no).

CONTACTS AND LOCATIONS:
Overall Officials: Paula Berstad, PhD, Principal Investigator — Norwegian Institute of Public Health
Locations (1):
- Norwegian Institute of Public Health, Oslo, Norway